CLINICAL TRIAL: NCT02570308
Title: A Phase I/II Open-label, Multi-center Study of the Safety and Efficacy of IMCgp100 Using the Intra-patient Escalation Dosing Regimen in Patients With Advanced Uveal Melanoma
Brief Title: A Study of the Intra-Patient Escalation Dosing Regimen With IMCgp100 in Patients With Advanced Uveal Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMCgp100-102
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Results first posted 2021-09-01 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Uveal Melanoma
Keywords: Tebentafusp; IMCgp100; gp100; metastatic melanoma; ImmTAC; Immunotherapy; Bispecific T cell receptor fusion protein; Immune mobilizing monoclonal T cell receptor; against cancer; UM; mUM; Kimmtrak
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Dose escalation (Experimental): Dose escalation cohorts of the intra-patient escalation regimen.
  Interventions: Drug: IMCgp100
- Dose expansion (Experimental): Dose expansion cohort with the recommended phase 2 dose of the intra-patient dose escalation regimen.
  Interventions: Drug: IMCgp100

INTERVENTIONS:
Drug: IMCgp100 — Bispecific soluble HLA-A2 restricted gp100-specific T-cell receptor fused to anti-CD3
  Other Names: Tebentafusp; Kimmtrak

SUMMARY:
IMCgp100-102 is a Phase I/II study of the weekly intra-patient escalation dose regimen with IMCgp100 as a single agent in participants with metastatic uveal melanoma (mUM). According to this regimen, all participants in the trial received 2 weekly doses of IMCgp100 at a dose level below the identified weekly recommended Phase II dose (RP2D-QW) and then a dose escalation commenced at the third weekly dose at C1D15. The Phase I testing of the intra-patient escalation dosing regimen is designed to achieve a higher exposure and maximal plasma concentration of IMCgp100 after doses at Cycle 1 Day 15 (C1D15) and thereafter.

DETAILED DESCRIPTION:
This is a Phase I/II clinical study of IMCgp100 in participants with advanced uveal melanoma.

This is a Phase I/II study of IMCgp100 administered on a weekly basis with an intra-patient escalation dosing regimen. The intra-patient escalation occurred at the third weekly dose on Cycle 1 Day 15 (C1D15). According to this regimen, all participants in the trial received 2 weekly doses of IMCgp100 at a dose level below the identified weekly recommended Phase II dose (RP2D-QW), and then a dose escalation commenced at the third weekly dose at C1D15 with the goal to achieve a long-term dosing regimen at a dose higher than that identified for the weekly dosing regimen (RP2D-QW). The dose escalation identified the intra-patient escalation regimen (RP2D-IE).

The Phase I portion of the study was a standard 3+3 dose escalation design.The recommended Phase II dose of the intra-patient escalation dose regimen (RP2D-IE) was identified and expansion cohorts in metastatic uveal melanoma was accrued based on prior therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants age ≥ 18 years of age at the time of informed consent.
2. Ability to provide and understand written informed consent prior to any study procedures.
3. Histologically or cytologically confirmed diagnosis of metastatic uveal melanoma (mUM).
4. Surgically sterile participants or participants of child-bearing potential who agree to use highly effective methods of contraception during study dosing and for 6 months after last dose of study drug.
5. Human leukocyte antigen (HLA)-A*0201 positive.
6. ECOG Performance Status of 0 or 1 at Screening.
7. Phase 2 will include participants with previously treated uveal melanoma in the metastatic setting.

Exclusion Criteria:

1. Presence of symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases that require doses of corticosteroids.
2. History of severe hypersensitivity reactions to other biologic drugs or monoclonal antibodies.
3. Participants with any out-of-range laboratory values.
4. Clinically significant cardiac disease or impaired cardiac function.
5. Active infection requiring systemic antibiotic therapy.
6. Known history of HIV infection.
7. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol.
8. Participants receiving systemic treatment with systemic steroid therapy or any other immunosuppressive medication at any dose level that would interfere with the action of the study drugs in the opinion of the investigator.
9. Malignant disease, other than that being treated in this study.
10. Any medical condition that would, in the investigator's judgment, prevent participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.
11. Presence of NCI CTCAE ≥ grade 2 toxicity (except alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ NCI CTCAE grade 3) due to prior cancer therapy.
12. Pregnant, likely to become pregnant, or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (17):
  - University California, San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - W LA Office, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Miami Hospital Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Washington University, School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center - The New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Hospital, New York, New York
  - Dean A. Mcgee Eye Institute, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Thomas Jefferson University Medical Oncology Clinic, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Health, Temple, Texas
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Germany (2):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
- Spain (4):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (2):
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral, Merseyside
  - Mount Vernon Cancer Centre, Northwood, Middlesex

REFERENCES:
- [Derived] Carvajal RD, Butler MO, Shoushtari AN, Hassel JC, Ikeguchi A, Hernandez-Aya L, Nathan P, Hamid O, Piulats JM, Rioth M, Johnson DB, Luke JJ, Espinosa E, Leyvraz S, Collins L, Goodall HM, Ranade K, Holland C, Abdullah SE, Sacco JJ, Sato T. Clinical and molecular response to tebentafusp in previously treated patients with metastatic uveal melanoma: a phase 2 trial. Nat Med. 2022 Nov;28(11):2364-2373. doi: 10.1038/s41591-022-02015-7. Epub 2022 Oct 13. PMID 36229663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 169 participants screened, 146 participants met the inclusion/exclusion criteria and were enrolled across 26 study centers in 5 countries.
Pre-assignment Details: The data cut-off date for this analysis was on 20 Mar 2020. The first patient was enrolled on 29 Feb 2016 in the Phase 1 dose escalation cohorts and on 19 Jan 2017 in the Phase 2 dose expansion cohort.
Groups:
- Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 54 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
- Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 64 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
- Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 73 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
- Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp; Phase 2 Dose Expansion: 68 mcg Tebentafusp: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 68 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
Period: Overall Study
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp | Phase 2 Dose Expansion: 68 mcg Tebentafusp
Started | 3 | 6 | 4 | 6 | 127
Completed | 2 | 1 | 0 | 2 | 53
Not Completed | 1 | 5 | 4 | 4 | 74
Not completed — Death | 1 | 5 | 4 | 4 | 69
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised all participants assigned to study drug and who received at least 1 full or partial dose of tebentafusp.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp | Phase 2 Dose Expansion: 68 mcg Tebentafusp | Total
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 127 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (6.03) | 54.7 (11.99) | 56.5 (18.41) | 55.8 (9.24) | 61.0 (10.93) | 60.4 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 64 | 74
  Male | 1 | 3 | 2 | 3 | 63 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 6 | 4 | 6 | 126 | 145
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT) in Phase 1
Description: Number of participants with a dose limiting toxicity, defined as an adverse event (AE) or abnormal laboratory value assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle of treatment and meets any of the pre-specified criteria.
Time Frame: Up to 49 months
Population: The Safety Analysis Set (SAS) included all participants who received at least 1 full or partial dose of tebentafusp.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp
Number analyzed (Participants) | 3 | 6 | 4 | 6
Participants | 0 | 1 | 2 | 0

2. Primary Outcome: Objective Response Rate in Phase 2
Description: Objective response rate (ORR) is defined as the percentage of participants with measurable disease with at least 1 visit response of complete response (CR) or partial response (PR) that is confirmed at least 4 weeks later, as defined in RECIST v.1.1 and assessed by an independent central review (ICR). The denominator in the calculation of the ORR is the number of participants in the full analysis set with measurable disease at baseline.
Time Frame: Up to 38 months
Population: The Full Analysis Set (FAS) included all participants who received at least 1 full or partial dose of tebentafusp.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Dose Expansion: 68 mcg Tebentafusp
Number analyzed (Participants) | 127
Percentage of participants | 4.7 [1.8 to 10.0]

3. Secondary Outcome: Objective Response Rate in Phase 1
Description: ORR is defined as the percentage of participants with measurable disease with at least 1 visit response of CR or PR that is confirmed at least 4 weeks later, as defined in RECIST v.1.1 and assessed by an investigator. The denominator in the calculation of the ORR is the number of participants in the full analysis set with measurable disease at baseline.
Time Frame: Up to 49 months
Population: The Full Analysis Set (FAS) included all participants who received at least 1 full or partial dose of tebentafusp. The analysis was pre-specified to be a pooled analysis of all Phase 1 cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 1 Dose Escalation: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) doses per cohort administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
Arm/Group | Phase 1 Dose Escalation
Number analyzed (Participants) | 19
Percentage of participants | 15.8 [3.4 to 39.6]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time in months from first dose of study drug until the date of disease progression or death (by any cause in the absence of disease progression) as assessed by RECIST v1.1 by the investigator for Phase 1 and ICR for Phase 2.
Time Frame: Up to 49 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2 Dose Expansion: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 68 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days).
Arm/Group | Phase 1 Dose Escalation | Phase 2 Dose Expansion
Number analyzed (Participants) | 19 | 127
Months | 7.4 [1.2 to 14.8] | 2.8 [2.0 to 3.7]

5. Secondary Outcome: Disease Control Rate
Description: Disease control rate (DCR) is defined as the percentage of participants with a best overall response of CR or PR or stable disease (SD) recorded at least 24 weeks (± 1 week) after commencement of study drug and prior to any progressive disease (PD) event, as assessed by RECIST v1.1 by the investigator for Phase 1 and ICR for Phase 2.
Time Frame: 24 weeks
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1 Dose Escalation | Phase 2 Dose Expansion
Number analyzed (Participants) | 19 | 127
Percentage of participants | 47.4 [24.4 to 71.1] | 22.8 [15.9 to 31.1]

6. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) is defined as the time in months from the date of first documented objective response (CR or PR) until the date of documented disease progression or death by any cause in the absence of disease progression as assessed by RECIST v1.1 by the investigator for Phase 1 and ICR for Phase 2.
Time Frame: Up to 49 months
Population: The analysis population included all participants who received at least 1 full or partial dose of tebentafusp and who achieved a response. The analysis was pre-specified to be a pooled analysis of all Phase 1 cohort participants (irrespective of dose); therefore, data by individual dose were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 Dose Escalation | Phase 2 Dose Expansion
Number analyzed (Participants) | 3 | 6
Months | 7.425 [3.713 to NA] — Not calculable because an insufficient number of participants reached the event at the final time point for assessment | 8.706 [5.552 to 24.542]

7. Secondary Outcome: Time to Response
Description: Time to response (TTR) is defined as the time in months from the date of first dose of study drug until the date of first documented objective response as assessed by RECIST v1.1 by the investigator for Phase 1 and ICR for Phase 2.
Time Frame: Up to 49 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Phase 1 Dose Escalation | Phase 2 Dose Expansion
Number analyzed (Participants) | 3 | 6
Months | 5.5 (1.8) | 7.0 (6.9)

8. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time in months from the date of first dose of study drug until death due to any cause in general.
Time Frame: Up to 49 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1 Dose Escalation | Phase 2 Dose Expansion
Number analyzed (Participants) | 19 | 127
Months | 29.6 [10.9 to 42.2] | 16.8 [12.9 to 21.3]

9. Secondary Outcome: Minor Response Rate
Description: Rate of minor response (or better) is defined as the proportion of participants with a confirmed CR, PR, or minor response (MinR) as assessed by RECIST v1.1 by the investigator for Phase 1 or ICR for Phase 2, where MinR is a reduction from baseline in sum of diameters between 10%-29%. The sum of diameters is defined as per RECIST v1.1 as the sum of longest diameters or short axis of target lesions (mm).
Time Frame: Up to 49 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1 Dose Escalation | Phase 2 Dose Expansion
Number analyzed (Participants) | 19 | 127
Percentage of participants | 26.3 [9.1 to 51.2] | 11.0 [6.2 to 17.8]

10. Secondary Outcome: Number of Participants With Treatment Dose Interruptions or Reductions
Description: Tolerability of study treatment was assessed by summarizing the number of participants with dose interruptions or reductions that occurred during the treatment period.
Time Frame: Up to 49 months
Population: The Safety Analysis Set (SAS) included all participants who received at least 1 full or partial dose of tebentafusp.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Escalation Cohort 2: 73 mcg Tebentafusp: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 73 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
- Phase 1 Dose Escalation Cohort 2: 68 mcg Tebentafusp; Phase 2 Dose Expansion: Fixed low doses of 20 mcg tebentafusp at Cycle 1 Day 1 (C1D1) and 30 mcg at Cycle 1 Day 8 (C1D8), followed by weekly (QW) 68 mcg dose administered intravenously at Cycle 1 Day 15 (C1D15) and beyond (each cycle is 28 days)
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 68 mcg Tebentafusp | Phase 2 Dose Expansion
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 127
Participants | 2 | 4 | 3 | 4 | 49

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Tebentafusp
Description: The AUC was determined in in dose escalation cohorts.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: predose, end of infusion, and 4 and 8 hours postdose
Population: All participants who received at least 1 full or partial dose of tebentafusp and with detectable serum concentrations are included.
Measure: Geometric Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp
Number analyzed (Participants) | 3 | 6 | 4 | 6
hr*pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 6
  Cycle 1 Day 1 | 28550 (27.0) | 36530 (23.3) | 32920 (18.2) | 33030 (16.5)
  Cycle 1 Day 15 | 81310 (33.7) | 98660 (34.8) | 106800 (11.6) | 109800 (23.3)

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Tebentafusp
Description: The Cmax is determined in dose escalation cohorts.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: predose, end of infusion, and 4 and 8 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp
Number analyzed (Participants) | 3 | 6 | 4 | 6
pg/mL
  Cycle 1 Day 1 | 3050 (15.1) | 3294 (22.7) | 3041 (21.7) | 3640 (23.3)
  Cycle 1 Day 15 | 8885 (17.2) | 9523 (23.0) | 11300 (11.7) | 11520 (25.8)

13. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Tebentafusp
Description: The Tmax of tebentafusp is determined in dose escalation cohorts.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: predose, end of infusion, and 4 and 8 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp
Number analyzed (Participants) | 3 | 6 | 4 | 6
Hours
  Cycle 1 Day 1 | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50]
  Cycle 1 Day 15 | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50]

14. Secondary Outcome: Apparent Terminal Plasma Half-life (t½) of Tebentafusp
Description: The t½ of tebentafusp is reported in dose escalation cohorts.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: predose, end of infusion, and 4 and 8 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp
Number analyzed (Participants) | 3 | 6 | 4 | 6
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 6
  Cycle 1 Day 1 | 6.635 [5.40 to 6.67] | 7.591 [6.03 to 11.3] | 6.442 [5.82 to 7.63] | 6.273 [5.59 to 10.1]
  Cycle 1 Day 15 | 6.897 [6.78 to 8.03] | 7.532 [6.57 to 10.5] | 7.519 [6.36 to 9.24] | 7.488 [5.70 to 11.9]

15. Secondary Outcome: Percentage of Participants With Anti-IMCgp100 Antibody Formation
Description: Overall antidrug antibody (ADA) is presented as number of ADA-positive participants relative to total number of participants with evaluable ADA results in each cohort
Time Frame: Up to 49 months
Population: The Full Analysis Set (FAS) included all participants who received at least 1 full or partial dose of tebentafusp and with evaluable data; two participants were excluded from ADA evaluation due to lack of sampling after dosing.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp | Phase 2 Dose Expansion: 68 mcg Tebentafusp
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 125
Percentage of participants | 66.7 | 16.7 | 25.0 | 33.3 | 33.6

ADVERSE EVENTS:
Time Frame: Up to 49 months
Description: Adverse events (AEs) are defined as treatment-emergent AEs that started or worsened after the first dose of study drug and within 90 days after the last dose.
Arm/Group | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp | Phase 2 Dose Expansion: 68 mcg Tebentafusp
All-Cause Mortality (participants affected / at risk) | 1/3 | 5/6 | 4/4 | 4/6 | 69/127
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 3/4 | 3/6 | 42/127
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 4/4 | 6/6 | 127/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp (N=3) | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp (N=6) | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp (N=4) | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp (N=6) | Phase 2 Dose Expansion: 68 mcg Tebentafusp (N=127)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 9 (11)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ system dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
General physical condition decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Rash generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infarction (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation Cohort 1: 54 mcg Tebentafusp (N=3) | Phase 1 Dose Escalation Cohort 2: 64 mcg Tebentafusp (N=6) | Phase 1 Dose Escalation Cohort 3: 73 mcg Tebentafusp (N=4) | Phase 1 Dose Escalation Cohort 4: 68 mcg Tebentafusp (N=6) | Phase 2 Dose Expansion: 68 mcg Tebentafusp (N=127)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 17 (21)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 12 (15)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 15 (22)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otorrhea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parasthesia ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dry eye (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 9 (12)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eyelash hypopigmentation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Ocular hyperemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Periorbital edema (Eye disorders) | 1 (2) | 4 (13) | 3 (9) | 4 (9) | 34 (69)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (7)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 14 (16)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (9) | 3 (7) | 2 (7) | 45 (71)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 26 (38)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (5) | 3 (4) | 30 (45)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (13) | 3 (7) | 4 (11) | 33 (50)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (5) | 15 (21)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 16 (23)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (7) | 5 (21) | 4 (18) | 5 (14) | 86 (247)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (13) | 3 (5) | 4 (11) | 52 (141)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (20)
Chest pain (General disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 2 (8) | 3 (14) | 4 (48) | 5 (20) | 84 (282)
Face edema (General disorders) | 0 (0) | 2 (2) | 1 (4) | 2 (4) | 15 (32)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (9) | 5 (16) | 4 (6) | 6 (21) | 78 (134)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (7) | 2 (21) | 1 (1) | 23 (49)
Infusion site hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 9 (10)
Nodule (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 4 (4)
Edema peripheral (General disorders) | 3 (3) | 5 (9) | 3 (12) | 5 (7) | 44 (86)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (15) | 6 (16) | 3 (16) | 6 (21) | 103 (417)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 7 (10)
Hyperbilirubinemia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 10 (16)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (45)
Diverticulitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localized infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (18)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (3) | 1 (2) | 0 (0) | 11 (16)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 16 (18)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 3 (11) | 1 (5) | 1 (1) | 5 (11)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 2 (3)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 19 (33)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (6) | 2 (3) | 0 (0) | 23 (36)
Blood alklaline phosphatase increased (Investigations) | 0 (0) | 2 (5) | 0 (0) | 3 (3) | 13 (19)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 12 (19)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 20 (20)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (13)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (3) | 32 (45)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 10 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 14 (24)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 14 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 3 (6) | 1 (2) | 33 (45)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 5 (24) | 4 (5) | 2 (4) | 41 (57)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (8) | 1 (5) | 1 (3) | 23 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (19) | 3 (10) | 2 (3) | 19 (33)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (10) | 2 (2) | 1 (2) | 12 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (3) | 1 (2) | 11 (14)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 6 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (9) | 1 (5) | 0 (0) | 2 (2) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (4) | 0 (0) | 0 (0) | 8 (11)
Tumor inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (6) | 2 (2) | 4 (12) | 42 (91)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 2 (4) | 3 (3) | 21 (25)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (4) | 2 (3) | 1 (2) | 10 (15)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 12 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 7 (9)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 20 (23)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 13 (13)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (13)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (8) | 0 (0) | 5 (9) | 29 (49)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (4) | 2 (6) | 24 (34)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 13 (16)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (6) | 2 (4) | 1 (4) | 10 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 1 (3) | 1 (1) | 3 (4)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (4)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 4 (25) | 4 (18) | 6 (26) | 87 (206)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 2 (3) | 5 (9) | 52 (68)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 51 (121)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (4) | 2 (6) | 42 (88)
Hair color changes (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (7) | 34 (38)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (20) | 3 (19) | 2 (8) | 22 (33)
Rash generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 30 (63)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (4) | 25 (31)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 28 (32)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 21 (22)
Generalized erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (4) | 0 (0) | 20 (59)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 22 (70)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 12 (12)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (11) | 0 (0) | 1 (1) | 11 (15)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 11 (13)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (13)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (7)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 1 (12) | 1 (1) | 5 (18)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (9) | 2 (15) | 2 (5) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Ephelides (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Miiaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (8) | 4 (5) | 2 (4) | 5 (10) | 53 (115)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 18 (53)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 14 (26)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT02570308/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02570308/SAP_001.pdf